CLINICAL TRIAL: NCT00777543
Title: The Effect of Pre-treatment of Bran on the Bioavailability of Ferulic Acid and Other Bioactive Compounds From Wholegrain Breads Enriched in Bran
Brief Title: Increasing Ferulic Acid Bioavailability in Bran
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 08-3-079; NL26116.068.08
Record Dates: First submitted 2008-10-16; First posted 2008-10-22 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2009-11

CONDITIONS: Healthy Males
Keywords: Bioavailability; Ferulic acid; Phenolic compounds; Colonic metabolites; Immunomodulatory effects; No disease
MeSH Terms: interventions — ferulic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): The control is the wholegrain bread enriched with bran that has not been pretreated.
  Interventions: Other: ferulic acid; Dietary Supplement: wholegrain bread
- Treated bran bread (Experimental): This is a wholegrain bread enriched with bran that has been pretreated with food-grade enzymes and yeast fermentation
  Interventions: Other: ferulic acid; Dietary Supplement: Treated bran bread

INTERVENTIONS:
Other: ferulic acid — Ferulic acid is naturally contained in wholegrain bread. Bran is the main source of ferulic acid while is low in white flour. Ferulic acid is mainly covalently bound to fiber and low bioaccessible. The bran is pretreated to increase the bioavailability of ferulic acid by increasing the free ferulic acid released from the food matrix.
  Other Names: Wholegrain bread; Bran; 4-hydroxy-3-methoxycinnamic acid
Dietary Supplement: Treated bran bread — This is a wholegrain bread enriched with bran that has been pretreated with food-grade enzymes and yeast fermentation
  Arms: Treated bran bread
Dietary Supplement: wholegrain bread — The control is the wholegrain bread enriched with bran that has not been pretreated
  Arms: Control

SUMMARY:
The aim of the present study is to investigate the effect of pretreatment of bran on improving the bioavailability of ferulic acid in wholegrain breads containing bran. As secondary endpoints we will investigate the changes in plasmatic antioxidant capacity, anti-inflammatory effects, colonic metabolites from ferulic acid and short chain fatty acids (SCFA).

DETAILED DESCRIPTION:
Rationale: Whole grain consumption has been associated with a lower risk of developing metabolic syndrome, cardiovascular disease, type 2 diabetes and some type of cancers. Whole grain is a good source of antioxidant compounds such as ferulic acid, which has been considered its major antioxidant. Ferulic acid is also the major phenolic compound in wheat grain, it is mainly located in the bran, more precisely in the cell walls of the aleurone layer and overall bran layers. Most of the ferulic acid is covalently bound to the indigestible cell wall polysaccharides, which limits the bioavailability of ferulic acid from cereal products to the merely form of free ferulic acid.

Processing possibilities in the development of cereal products might be used to optimize the bioavailability of ferulic acid in humans and the possible health effect of the wholegrain product.

An innovative processing in bread making has been developed. The processing consisted of pretreatments of the bran with an enzymatic mixture and yeast fermentation before its incorporation into the dough. The impact on the in vitro assessed bioavailability of ferulic acid was a 5-fold increase over the normal bran enriched wholegrain bread in a gastrointestinal model. Therefore in our study we will compare the kinetics and total bioavailability of ferulic acid from wholegrain breads enriched in native or pretreated bran. Furthermore, the colonic metabolism of ferulic acid and overall major colonic metabolites such as short chain fatty acids (SCFA) will be studied. Finally, total antioxidant capacity and ex vivo inflammatory responses will be investigated in order to determine the effect of the pretreatment of on the immunomodulatory properties of bran.

Objective: The aim of the present study is to investigate the effect of pretreatment of bran on improving the bioavailability of ferulic acid. As secondary endpoints we will investigate the changes in plasmatic antioxidant capacity, anti-inflammatory effects, colonic metabolites from ferulic acid and short chain fatty acids (SCFA).

Study design: Blind, cross-over, randomised design. Wash-out period of one week. Three days of low antioxidant diet. Standardised meal low in phenolic and antioxidant compounds will be consumed the evening before the trial.

Study population: Healthy male volunteers, > 18 yr old, BMI between 20 and 30. Intervention: Consumption of 300 g of wholegrain enriched with native or pretreated bran.

Main study parameters/endpoints: Ferulic acid and other phenolic acids (sinapic acid, p-coumaric acid), total antioxidant capacity, anti-inflammatory effects, colonic metabolites derived from ferulic acid and SCFA.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Each volunteer will participate in the study on two separate occasions (each test will take approximately 24 hours). Blood will be drawn at different time points via a catheter (in total 156 ml per test-day) and a 24-hour urine sample will be collected. Participants are asked to consume a standardised meal the evening before each of the two test-days and the evening of the intervention day. Volunteers are instructed not to consume any wholegrain or bran containing products, nuts and seeds, antioxidant supplements or beverages high in phenolic compounds or any phenolic rich food for 3 days before each of the three trials. Subjects are asked to record their food intake for 3 days before each of the trials. All the ingredients used in the bread baking are safe for human consumption. The bread is consumed once at the beginning of the test. The volunteers will not benefit from the study. The major risk of the study is the amount of blood take from the volunteer and this risk is limited.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age > 18
* 20 < BMI < 30

Exclusion Criteria:

* Use of any medication
* Smoking
* Consumption of 3 or more glasses of alcoholic drinks per day
* Donation of more than 500 ml blood (<6 months prior to the start of the study)
* Vegetarian lifestyle (because the standardised meal contains meat)
* Allergic reaction to some component in cereals e.g. celiac subjects

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Ferulic acid is measured in plasma to determine maximal concentration (Cmax), time-point of Cmax (tmax) and area under the curve (AUC). Ferulic acid is also measured in 24-hour urine sample to determine its excretion. | 24 h

SECONDARY OUTCOMES:
Colonic metabolites derived from ferulic acid, short chain fatty acids and antioxidant capacity are measured in plasma to determine their relation with the plasma levels of ferulic acid. Cytokines will be measured in ex vivo LPS stimulated blood. | 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Aalt Bast, Professor, Principal Investigator — Universit of Maastricht
Locations (1):
- University of Maastricht, Maastricht, Netherlands